CLINICAL TRIAL: NCT02303054
Title: Magnetic Resonance (MR)-US Fusion Biopsy-Guided Focal Bipolar Radio-Frequency Ablation of the Prostate in Men With Localized Prostate Cancer (FUSAblate Trial)
Brief Title: MRI-Targeted Focal Ablation of the Prostate in Men With Prostate Cancer
Acronym: FUSAblate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Trod Medical N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-00903
Record Dates: First submitted 2014-11-08; First posted 2014-11-27 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Focal Ablation; MRI-US Fusion Biopsy; Focal Therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bipolar Radiofrequency Focal Ablation (Experimental): Men identified as having suspicious regions on an Prostatic multi-parametric MRI (mpMRI) of the prostate will be considered for enrollment. If followed by a positive MRI-US targeted biopsy of the prostate, men who be offered enrollment into the study. All men enrolled in the study will undergo bipolar radiofrequency ablation. Efficacy will be assessed through MRI-US biopsy after focal bipolar RFA.
  Interventions: Procedure: Bipolar Radiofrequency Focal Ablation

INTERVENTIONS:
Procedure: Bipolar Radiofrequency Focal Ablation — Men identified as having suspicious regions on a pre-biopsy mpMRI will be considered for enrollment. Following an MRI-US targeted biopsy of the prostate, men testing positive will be eligible for enrollment. All men enrolled in the study will undergo focal radiofrequency ablation and evaluated in follow-up.

SUMMARY:
This is a prospective single center trial to examine the rate of negative biopsy result and quality of life after focal ablation by radiofrequency energy. The primary evaluation involves assessing the rate of negative biopsy result using MR-US fusion biopsy six months after focal ablation of the prostate. Urinary and sexual quality of life will be assessed through validated measures. The hypothesis of our study is that focal ablative therapy will result in a greater likelihood of negative biopsy on followup biopsy than that observed in men who elect not to undergo therapy.

ELIGIBILITY:
Inclusion Criteria:

Subject Population:

* Men 40-80 years of age
* Diagnosis of adenocarcinoma of the prostate, confirmed by TransRectal Ultrasound (TRUS) biopsy
* No prior treatment for prostate cancer
* Prostate Cancer Clinical Stage T1c
* Prostate-specific antigen (PSA)<10 ng/ml (this will be the PSA level prompting the initial prostate biopsy)
* Declined all standard treatment options

Pre-enrollment biopsy parameters:

* Minimum of 12 biopsy cores
* Gleason 6 (3+3) or 7 (3+4)

Final enrollment biopsy parameters after fusion biopsy:

* 12 standard biopsy cores plus targeted regions based upon MRI
* Gleason 6 (3+3) or 7 (3+4)
* No demonstrated cancer diameter >1.2 cm

Exclusion Criteria:

* Histology other than adenocarcinoma
* Biopsy does not meet inclusion criteria
* History of transurethral resection of prostate (TURP) or other similar procedures transurethral microwave therapy (TUMT), transurethral needle ablation (TUNA)
* History of prior pelvic radiation
* Men who have received any hormonal manipulation (antiandrogens; luteinizing hormone-releasing hormone (LHRH)-agonist; 5-alpha-reductase inhibitors) within the previous 12 months
* Contraindication for Multiparametric-MRI

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of Subjects Resulting in Negative Biopsy as a Measure of Efficacy | 6 months after focal bipolar radiofrequency ablation (RFA)
  The primary endpoint of the trial will be assessed at 6 months after focal bipolar RFA by repeat mp-MRI imaging and fusion biopsy. Treatment efficacy, defined as a negative, will be determined by the results of the MRI-US targeted biopsy that will include regions treated by focal bipolar RFA.

SECONDARY OUTCOMES:
International Prostate Symptom Score to Measure Quality of Life Post Focal Ablation | 1 week; 2 week; 1 month; 3 months; 6 months
  Participants will be asked to complete international prostate symptom score (IPSS) questionnaires at each time frame to determine any baseline changes from voiding symptoms following focal RFA
Expanded Prostate Cancer Index Composite (EPIC) Score to Measure Quality of Life Post Focal Ablation | 1 week; 2 week; 1 month; 3 months; 6 months
  Participants will be asked to complete EPIC questionnaires at each time frame to evaluate any baseline changes in patient function and bother following focal RFA
International Index of Erectile Function questionnaires Score (IEFF) to Measure Quality of Life Post Focal Ablation | 1 week; 2 week; 1 month; 3 months; 6 months
  Participants will be asked to complete International Index of Erectile Function (IIEF) - 15 questionnaires at each time frame to evaluate any baseline changes in erectile function following focal RFA
Short Form - 12 (SF-12) to Measure Quality of Life Post Focal Ablation | 1 week; 2 week; 1 month; 3 months; 6 months
  Participants will be asked to complete SF-12 questionnaires at each time frame to evaluate any baseline changes in functional health and well-being

CONTACTS AND LOCATIONS:
Overall Officials: Samir S Taneja, MD, Principal Investigator — NYU Langone Health
Locations (1):
- Smilow Comprehensive Prostate Cancer Center, New York, New York, United States